CLINICAL TRIAL: NCT06624488
Title: The Relationship Between Brain Injury Biomarkers in Cerebrospinal Fluid and Blood of Patients After Cardiac Arrest and Prognosis.
Status: Recruiting | Type: Observational
Sponsor: Tang Ziren (Other)
Responsible Party: Sponsor-Investigator, Tang Ziren, Professor, Capital Medical University
Organization: Capital Medical University (Other)
Other Study IDs: 2023-1-10-3
Record Dates: First submitted 2024-09-30; First posted 2024-10-03 (Actual); Last update posted 2025-02-21 (Actual); Status verified 2025-02

CONDITIONS: Cardiac Arrest (CA); Brain Injuries, Acute
Keywords: cardiac arrest; brain injury; cerebrospinal fluid; biomarkers
MeSH Terms: conditions — Heart Arrest; Brain Injuries

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This study is a single-center, prospective, observational study. After successful cardiopulmonary resuscitation for patients with cardiac arrest, they will be transferred to the emergency intensive care unit for further standardized targeted temperature management. When evaluating that the patient meets the indications for lumbar puncture and there are no contraindications for lumbar puncture, lumbar puncture examinations will be completed immediately after return of spontaneous circulation (ROSC), at 24 hours of hypothermia, at 72 hours of hypothermia, and after rewarming. Routine cerebrospinal fluid examinations such as cerebrospinal fluid routine, cerebrospinal fluid biochemistry, and cerebrospinal fluid lactate will be sent for inspection. At the same time, 6 ml of cerebrospinal fluid will be retained and stored in a refrigerator at -80°C. After sample collection is completed, enzyme-linked immunosorbent assay (ELISA) will be used to detect markers such as NSE, HCH-L1, NFL, tau, MBP, GFAP, and S100β. While performing the lumbar puncture examination, peripheral blood will be collected. After centrifugation for 10 minutes (4000 revolutions), serum will be retained and stored in a refrigerator at -80°C to complete the examination of the above markers. After 3 months, the patient's neurological function prognosis will be followed up according to the Pittsburgh Cerebral Performance Category (CPC) scale.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years old.
* Still lack of directive movements after restoration of spontaneous circulation through cardiopulmonary resuscitation.
* Advanced life support and targeted temperature management are carried out within 6 hours after return of spontaneous circulation (ROSC).

Exclusion Criteria:

* Patients with contraindications for lumbar puncture (severe cerebral edema indicated by brain imaging, disappearance of basal cisterns or occult intracranial mass lesions, receiving antiplatelet and anticoagulant therapy, and those with coagulation disorders).
* Pregnant patients.
* Patients with concomitant traumatic brain injury, stroke, cerebral hemorrhage and other diseases.
* Patients whose families do not agree to be enrolled.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients after successful cardiopulmonary resuscitation (CPR) were transferred to the emergency intensive care unit for further standardized management
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2023-01-01 (Actual); Primary Completion 2025-04-01 (Estimated); Study Completion 2025-05-01 (Estimated)

PRIMARY OUTCOMES:
Neurologic prognosis | 3 months
  Patients will be followed up for neurologic prognosis according to the Pittsburgh Cerebral Performance Category (CPC) scale at 3 months after disease onset.The CPC score ranges from 1 to 5, with 1 indicating good performance, 2 indicating moderate disability, 3 indicating severe disability, 4 indicating vegetative state and 5 indicating brain death or death.

CONTACTS AND LOCATIONS:
Locations (1):
- Beijing chaoyang hospital, Beijing, China